CLINICAL TRIAL: NCT06333418
Title: The Effect of Virtual Rain Forest and Glass Waterfall on Satisfaction, Comfort, Anxiety, and Vital Signs Undergoing Colonoscopy
Brief Title: Effects of VR and Glass WF Colonoscopy
Acronym: VR/WN_colon
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Hasan Genç, Asistant Professor, Dicle University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: VR/WF
Record Dates: First submitted 2024-03-13; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Misadventure During Endoscopic Examination
Keywords: virtual reality; glass waterfall; satisfaction; comfort; colonoscopy
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Parallel Assignment experimental model using randomized pretest and posttest with control group
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Glasses (Experimental): Before the colonoscopy procedure, 360-degree VR video scenes will be watched to patients 30 minutes using VR head device.
  Interventions: Device: Virtual Reality Glasses Group
- Glass waterfall (Experimental): Before the colonoscopy procedure, patients will watch and listen 30 minutes a portative glass waterfall
  Interventions: Device: Glass waterfall
- control group (No Intervention): Patients of the control group, will not receive any intervention except for applied routine hospital colonoscopy procedures

INTERVENTIONS:
Device: Virtual Reality Glasses Group — Before the colonoscopy procedure, 360-degree VR video scenes will be watched to patients 30 minutes using VR head device.
  Arms: Virtual Reality Glasses
Device: Glass waterfall — Before the colonoscopy procedure, patients will watch and listen 30 minutes a portative glass waterfall
  Arms: Glass waterfall

SUMMARY:
Background: Today, colonoscopy is widely used in many diseases, especially in the screening and diagnosis of colorectal cancers. Colonoscopy is considered a procedure that disturbs the patient's comfort because it is a very invasive and painful procedure. Along with physical discomfort during the procedure, it triggers emotional disturbances such as fear, and anxiety in the patient.

Purpose: To examine the effect of virtual rain forest and glass waterfall on satisfaction, comfort, anxiety, and vital signs before colonoscopy Method: The population of the study consists of all patients who applied to Mardin Education and Research Hospital, Department of General Surgery, Endoscopy Unit and were scheduled for colonoscopy. The sample will be represented by 135 patients whose colonoscopy procedure is planned between the specified dates and who meet the criteria for inclusion in the sample. In calculating the sample of the study, power analysis was performed and it was found the effect size of 0.40, 95% power and 0.01% margin of error for this study, that a total of 135 individuals for the three groups and at 60 individuals for each group. G*Power, version 3.0.10 was used for statistical power analysis. The study group of 93 people to participate in the study will be divided into three equal groups in accordance with the random numbers table obtained the computer- based Research Randomizer program. Before the arthroscopy procedure, the patients included in the study will be randomly divided into three groups: 45 rain forest video VR group, 45 glass waterfall group and 45 control group. All participants in the study will first fill out a patient identification form containing patient demographic information.

DETAILED DESCRIPTION:
Background: Today, colonoscopy is widely used in many diseases, especially in the screening and diagnosis of colorectal cancers. Colonoscopy is considered a procedure that disturbs the patient's comfort because it is a very invasive and painful procedure. Along with physical discomfort during the procedure, it triggers emotional disturbances such as fear, and anxiety in the patient.

Purpose: To examine the effect of virtual rain forest and glass waterfall on satisfaction, comfort, anxiety, and vital signs before colonoscopy Method: The population of the study consists of all patients who will apply to Mardin Education and Research Hospital, Department of General Surgery, Endoscopy Unit and will be scheduled for colonoscopy. The sample will be represented by 135 patients whose colonoscopy procedure is planned between the specified dates and who meet the criteria for inclusion in the sample. In calculating the sample of the study, power analysis will be performed and it will be found the effect size of 0.40, 95% power and 0.01% margin of error for this study, that a total of 135 individuals for the three groups and at 60 individuals for each group. G*Power, version 3.0.10 was used for statistical power analysis. The study group of 93 people to participate in the study will be divided into three equal groups in accordance with the random numbers table obtained the computer- based Research Randomizer program. Before the arthroscopy procedure, the patients included in the study will be randomly divided into three groups: 45 rain forest video VR group, 45 glass waterfall group and 45 control group. All participants in the study will first fill out a patient identification form containing patient demographic information. Before the colonoscopy procedure, 360-degree VR rain forest video scenes will be watched 30 minutes using VR head device in virtual glasses group. Glass Water group, patients will watch and listen 30 minutes a portative glass waterfall

ELIGIBILITY:
Inclusion Criteria:

* 18 aged and over
* Written and verbal consent to participate in the study,
* Being conscious (person, place and time orientation),
* Undergoing colonoscopy for the first time

Exclusion Criteria:

* Having vision, hearing and communication problems
* Having any psychiatric and cognitive/mental mental health problems, disease (dementia, etc.),
* Diagnosed with visual, auditory and / or balance disorders,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2024-04-03 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-08 (Estimated)

PRIMARY OUTCOMES:
Patient Information Form | the fundamental characteristics of the patients will be filled in 40 minutes before the colonoscopy procedure
  This form, which will be created by the researcher; Patients' age, gender, education level, marital status, employment status, income level, chronic disease status, previous surgery, complaints about coming to the hospital, having knowledge about colonoscopy, whether they would prefer the current method if they need to have colonoscopy again, It consists of a total of 14 questions questioning the use of additional sedation and painkillers during the procedure
Visual Analogue Scale (VAS) | Change from Baseline Visual Analogue Scale in 50 minutes
  This scale developed by Price (1983) will be used in the research to determine the level of tolerance, comfort and satisfaction. It is a scale in which the distance between the two ends with a minimum value of 0 on one end and a maximum value of 10 on the other end is measured with a 10 cm ruler. In this context; The patient is explained that there are two endpoints and that he is free to mark any place between them that fits the severity of his pain.
  The distance between the beginning of "no comfort, tolerance and satisfaction" and this point marked by the patient is measured and recorded in centimeters. It has been shown that the VAS is a valid tool for the measurement of psychological and health variables such as pain and satisfaction, which is widely used in clinical studies
State and Trait Anxiety Scale (STAI) | Change from Baseline The State and Trait Anxiety Scale in 50 minutes
  It is a self-assessment questionnaire developed by Spielberger et al. and consists of short assessments. The STAI includes 40 four-point Likert-type items ranging from "None" to "Completely". The validity and reliability of the STAI in Turkey were established by Öner and Le Compte. The STAI includes two separate scales, the State Anxiety Score (SAS) and the Trait Anxiety Score (TAS). The SAS requires the person to describe how they feel at a certain moment and under certain conditions and to respond by taking into account their feelings about the situation they are in. On the other hand, the TAS requires the person to describe how they usually feel. Higher scores indicate increased anxiety level. In the Turkish validity and reliability study, Cronbach's alpha reliability coefficients were between 0.83 and 0.87 for the TAS and between 0.94 and 0.96 for the SAS.
The Patient Observation Form | Change from Baseline The Patient Observation Form in 50 minutes
  This form will be created by the researcher based on the literature review, the vital signs (pulse (min), respiratory rate (min), systolic blood pressure (mmHg), diastolic blood pressure (mmHg), and oxygen saturation values (%)) of the patients before and after the procedure will be recorded the form. Researcher will has a automatic blood pressure monitor and a probe device for recording vital signs in the endoscopy unit. While the patients' vital signs will being taken, a fully automatic blood pressure monitor will be used to measure blood pressure and pulse. To measure the respiratory rate, the patient placed his hand on his chest and his chest movements will be counted and recorded for one minute. Oxygen saturation level will be measured from the index finger with a probe device.Data will be collected by recording all vital measurement values on a single form. The form will similar to forms commonly used in nursing research for patient vital signs.
Pulse rate before colonoscopy procedure | Change from Baseline Pulse rate in 50 minutes
  60 to 100 beats per minute is normal. It will be recorded 40 minutes (pretest) and 10 minutes (posttest) before the gastroscopy procedure
Respiratory rate before colonoscopy procedure | Change from Baseline Respiratory rate in 50 minutes
  12 to 18 breaths per minute is normal. It will be recorded 40 minutes (pretest) and 10 minutes (posttest) before the gastroscopy procedure
Systolic and diastolic blood pressure before colonoscopy procedure | Change from Baseline Systolic and diastolic blood pressure in 50 minutes
  90/60 mm Hg to 120/80 mm Hg is normal. It will be recorded 40 minutes (pretest) and 10 minutes (posttest) before the gastroscopy procedure
Oxygen saturation values before colonoscopy procedure | Change from Baseline Oxygen saturation values in 50 minutes
  Normal oxygen saturation usually ranges from 95 to 100%. It will be recorded 40 minutes (pretest) and 10 minutes (posttest) before the gastroscopy procedure

CONTACTS AND LOCATIONS:
Overall Officials: Hasan GENC, PhD, Principal Investigator — Dicle University

IPD SHARING:
Plan to Share IPD: No
all IPD that underlie results in a publication

REFERENCES:
- [Background] Huang MY, Scharf S, Chan PY. Effects of immersive virtual reality therapy on intravenous patient-controlled sedation during orthopaedic surgery under regional anesthesia: A randomized controlled trial. PLoS One. 2020 Feb 24;15(2):e0229320. doi: 10.1371/journal.pone.0229320. eCollection 2020. PMID 32092098
- [Result] Sahin G, Basak T. The Effects of Intraoperative Progressive Muscle Relaxation and Virtual Reality Application on Anxiety, Vital Signs, and Satisfaction: A Randomized Controlled Trial. J Perianesth Nurs. 2020 Jun;35(3):269-276. doi: 10.1016/j.jopan.2019.11.002. Epub 2020 Mar 4. PMID 32146074
- [Result] Celebi D, Yilmaz E, Sahin ST, Baydur H. The effect of music therapy during colonoscopy on pain, anxiety and patient comfort: A randomized controlled trial. Complement Ther Clin Pract. 2020 Feb;38:101084. doi: 10.1016/j.ctcp.2019.101084. Epub 2019 Dec 23. PMID 32056820
- [Result] Umezawa S, Higurashi T, Uchiyama S, Sakai E, Ohkubo H, Endo H, Nonaka T, Nakajima A. Visual distraction alone for the improvement of colonoscopy-related pain and satisfaction. World J Gastroenterol. 2015 Apr 21;21(15):4707-14. doi: 10.3748/wjg.v21.i15.4707. PMID 25914482
- [Result] Veldhuijzen G, Klaassen NJM, Van Wezel RJA, Drenth JPH, Van Esch AA. Virtual reality distraction for patients to relieve pain and discomfort during colonoscopy. Endosc Int Open. 2020 Jul;8(7):E959-E966. doi: 10.1055/a-1178-9289. Epub 2020 Jun 30. PMID 32626819
- [Result] Ilkkaya NK, Ustun FE, Sener EB, Kaya C, Ustun YB, Koksal E, Kocamanoglu IS, Ozkan F. The effects of music, white noise, and ambient noise on sedation and anxiety in patients under spinal anesthesia during surgery. J Perianesth Nurs. 2014 Oct;29(5):418-26. doi: 10.1016/j.jopan.2014.05.008. PMID 25261145
- [Result] Rostom A, Ross ED, Dube C, Rutter MD, Lee T, Valori R, Bridges RJ, Pontifex D, Webbink V, Rees C, Brown C, Whetter DH, Kelsey SG, Hilsden RJ. Development and validation of a nurse-assessed patient comfort score for colonoscopy. Gastrointest Endosc. 2013 Feb;77(2):255-61. doi: 10.1016/j.gie.2012.10.003. PMID 23317691
- [Result] Dogan Yilmaz E, Unlusoy Dincer N. The Effects of Virtual Reality Glasses on Vital Signs and Anxiety in Patients Undergoing Colonoscopy: A Randomized Controlled Trial. Gastroenterol Nurs. 2023 Jul-Aug 01;46(4):318-328. doi: 10.1097/SGA.0000000000000733. Epub 2023 Jun 5. PMID 37278621